CLINICAL TRIAL: NCT04501796
Title: A Double-blind, Randomized, Placebo-controlled, Phase 1, Single-dose, Dose-escalating Trial of Long-acting Recombinant Human IL-7 (NT-I7) for COVID-19
Brief Title: A Trial of NT-I7 in COVID-19 (SPESELPIS)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was halted due to lack of patient population resulting in slow enrollment.
Sponsor: NeoImmuneTech (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIT-116 (SPESELPIS)
Record Dates: First submitted 2020-07-27; First posted 2020-08-06 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: COVID-19
Keywords: NT-I7 (efineptakin alfa, rhIL-7-hyFc); COVID-19
MeSH Terms: conditions — COVID-19 | interventions — efineptakin alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NT-I7 (Experimental): NT-I7 will be administered once by IM injection within 24 hours of baseline (day 0). The treatment course pursued in all enrolled participants will be a single dose. Dosing will be staggered with at least 72 hours between each study participant.
  Interventions: Drug: Double-Blind NT-I7
- Placebo (Placebo Comparator): Placebo will be administered once by IM injection within 24 hours of baseline (day 0). The treatment course pursued in all enrolled participants will be a single dose. Dosing will be staggered with at least 72 hours between each study participant.
  Interventions: Drug: Double-Blind Placebo

INTERVENTIONS:
Drug: Double-Blind NT-I7 — Administered by intramuscular (IM) injection
  Other Names: rhIL-7-hyFc; efineptakin alfa
  Arms: NT-I7
Drug: Double-Blind Placebo — Placebo
  Arms: Placebo

SUMMARY:
The main purposes of this study is to determine the following in participants with mild coronavirus disease 2019 (COVID-19):

* Safety of a single dose of NT-I7
* The immunological effects of NT-I7 on peripheral lymphocyte counts in COVID-19 patients.

DETAILED DESCRIPTION:
This is a multisite, double-blind, randomized, placebo-controlled, dose-escalating, phase 1 trial of NT-I7 with standard of care (SOC) versus placebo with SOC to evaluate the safety and efficacy of NT-I7 in adults with mild coronavirus disease 2019 (COVID-19). After determination of eligibility and baseline assessment, a single dose of the study agent (NT-I7 or placebo) will be administered after 1:1 randomization, along with SOC. Research blood collection will occur at baseline, days 3, 7, 14, 30, 60 and 90 days after administration. Primary and secondary evaluations will include assessment of adverse events (AEs), absolute lymphocyte count (ALC), and trajectory of other lymphocytes subsets: CD4, CD8, natural killer (NK), B, and mucosal-associated-invariant T (MAIT) cells. The final study visit will be at day 90 after the study agent administration. The investigators hypothesize that NT-I7 is safe for administration and preserves lymphocyte homeostasis in patients with mild COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must meet all of the following criteria to be included in the study:
* Laboratory-confirmed SARS-CoV-2 infection as determined by either a documented positive molecular assay/ other commercial or public health assay in any specimen collected < 5 days prior to screening or a documented positive molecular assay ≥ 5 days prior to screening and confirmed by polymerase chain reaction (PCR) at screening.
* Illness of any duration with oxygen saturation > 93% at room air, heart rate ≤ 100 beats per minute at rest, and no evidence of respiratory distress with respiration rate < 20 breaths per minute.
* Able to provide informed consent.
* Aged ≥ 19 and ≤ 75 years.
* Absolute Lymphocyte Count <1,500 lymphocytes/µL.
* Avoid becoming pregnant or impregnate a partner through 90 days after study agent administration. Females must agree to 2 methods of contraception, and males to at least one method of contraception.
* Not participate in any other clinical trial for an investigational therapy through day 30.

Exclusion Criteria:

* Moderate to severe hypoxic respiratory failure requiring supplemental oxygen at rest, mechanical ventilation, ECMO, or any other noninvasive ventilation modality.
* CRP >15 mg/L or D-dimer > 0.75 µg/mL.
* Estimated glomerular filtration rate (eGFR) < 40 mL/min/1.73m2, or requiring dialysis.
* AST/ALT > 3-times ULN, or total bilirubin > 1.5 times ULN (except if due to Gilbert's syndrome).
* Pregnancy or breastfeeding.
* Use of systemic corticosteroids or immunomodulant within 4 weeks prior to screening.
* Receipt of an investigational agent or investigational use of a licensed agent within 16 weeks prior to screening.
* HIV infection or underlying history of known or unknown primary or acquired immunodeficiency associated with lymphopenia and/or recurrent opportunistic infections.
* Autoimmune disease requiring systemic treatment EXCEPT for vitiligo or endocrine disease (such as diabetes, thyroid disease, and adrenal disease) controlled by replacement therapy.
* Malignancy requiring treatment 1 year prior to screening.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-11-27 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of a single dose of NT-I7 in a dose escalation fashion | Up to approximately 30 days
  Assessment of the number and severity of AEs possibly, probably, or definitely related to study drug evaluated at 7 and 30 days.

SECONDARY OUTCOMES:
Evaluate the immunological effects of NT-I7 cumulatively for all doses on peripheral lymphocyte counts in COVID-19 patients. | Up to approximately 30 days
  Assessment of the trajectory of ALC, CD4, CD8, NK, B, and MAIT cells measured at days 7, 14 and 30 after administration of NT-I7 or placebo compared to baseline values.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Nih/Niaid, Bethesda, Maryland
  - University of Nebraska Medical Center, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: No